CLINICAL TRIAL: NCT02113475
Title: A Patient Outcome Study After Pharmacomechanical Catheter-directed Thrombolysis and Standard Treatment for Venous Thrombosis
Brief Title: Venous Thrombectomy/Thrombolysis Outcome Registry
Acronym: VETTOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heart and Vascular Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PC14-1213-001
Record Dates: First submitted 2014-04-09; First posted 2014-04-14 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Deep Venous Thrombosis; Post Thrombotic Syndrome
Keywords: CDT; PCDT; DVT; PTS; Quality of Life
MeSH Terms: conditions — Venous Thrombosis; Postthrombotic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Deep Venous Thrombosis affects more than 350,000 individuals each year in the U.S.The Registry will track patient outcome and quality of life over 60 months for treatment with anticoagulation and elastic compression stockings and catheter-directed thrombolysis (CDT) in accordance with current treatment guidelines .

ELIGIBILITY:
Inclusion Criteria:

•Data obtained in line with good clinical practice, applicable laws and regulation

Exclusion Criteria:

-

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participating study centers will enroll patients and enter data in the web-based registry that include demographics, clinical features,
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2014-04; Primary Completion 2020-03 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Life, | 60 months

SECONDARY OUTCOMES:
Rate of Post-Thrombotic Syndrome | 60 Months

CONTACTS AND LOCATIONS:
Overall Officials: Uchenna N Onyeachom, Study Director — Heart and Vascular Outcomes Research Institute
Locations (1):
- Heart & Vascular Outcomes Research Institute, Beverly, Massachusetts, United States